CLINICAL TRIAL: NCT03241251
Title: Screening for Psychosocial Risk in Flemish Families of a Child With Cancer
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S60600
Record Dates: First submitted 2017-07-28; First posted 2017-08-07 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Pediatric Cancer
Keywords: psychosocial risk
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- parents children pediatric cancer: Screening questionnaire psychosocial risk factors
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — Questionnaire of psychosocial risk factors

SUMMARY:
The Psychosocial Assessment Tool (PAT) is an international used instrument for the screening for psychosocial risk factors in families of a child with cancer. This study want to investigate the validation and evaluation of the clinical value of the Flemish translation of the psychosocial assessment tool

DETAILED DESCRIPTION:
Psychosocial support of children having a diagnosis of cancer and their families is a crucial aspect of a qualitative treatment. Assessment of psychosocial needs is a first step in order to provide better and preventive psychosocial support. In Flanders, no instrument for screening of psychosocial needs is available. The Psychosocial Assessment Tool (PAT) is an international used instrument for the screening for psychosocial risk factors in families of a child with cancer. This study want to investigate the validation and evaluation of the clinical value of the Flemish translation of the PAT. Two large Flemish pediatric oncology centers will participate: University hospital Ghent (UZGent) and the University hospital in Leuven (UZLeuven). During a time period of 2.5 years families in which a child received a new diagnosis of a pediatric cancer will be invited to participate in this study. All subscales of the PAT will be validated by the use of standardized parent questionnaires measuring similar constructs: Inventory Social Reliance, Strengths and Difficulties Questionnaire, Hospital Anxiety and Depression Scale, Parenting Stress Index-short version and illness cognitions questionnaire, parent version. The usability of the PAT will be evaluated with the PAT-Netherlands Usability questionnaire. The clinical value will be evaluated by comparing the clinical judgment of psychosocial risk by the psychosocial team members of both centers with the scores on the PAT.

The proposed project is an important step to ameliorate psychosocial support in families with a child with a diagnosis of cancer in Flemish pediatric oncological centers.

ELIGIBILITY:
Inclusion Criteria:

* parents of all children and adolescents from 0-18 years that are diagnosed with cancer

Exclusion Criteria:

* no knowledge of Dutch language

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: parents of all children and adolescents from 0-18 years that are diagnosed with cancer
Sampling Method: Non-Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2022-09-08 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
validation of PAT questionnaire | baseline assessment at diagnosis
  The PAT validation will be performed by correlating PAT scores with validated questionnaires measuring similar constructs as the PAT. These questionnaires are Inventory social reliance, strengths and difficulties questionnaire , hospital anxiety and depression scale, parenting stress index -short version and illness cognition questionnaire parent version.

SECONDARY OUTCOMES:
clinical value of questionnaire | baseline assessment at diagnosis
  a risk estimation of psychosocial risk by psychosocial team after diagnosis, but blinded to PAT scores, will be compared with PAT scores

CONTACTS AND LOCATIONS:
Overall Officials: Jurgen Lemiere, PhD, Study Director — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium